CLINICAL TRIAL: NCT02498522
Title: Effect of Metformin on Early Pregnancy Loss in Pregnant Women With Polycystic Ovarian Syndrome
Acronym: MIP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Islam Dabbous, doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Metformin in pregnancy
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin arm (Experimental): 83 patients will continue metformin until end of 1st trimester (14 weeks gestation)
  Interventions: Drug: Metformin
- control arm (Placebo Comparator): 83 patients will stop metformin at diagnosis of pregnancy ( 5-6 weeks gestation)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 83 patients will continue metformin until end of 1st trimester
  Other Names: cidophage

SUMMARY:
The aim of this work is to study the effect of metformin use for reducing early pregnancy loss in pregnant patients with Polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in women of reproductive age. PCOS produces symptoms in approximately 5 to 10% of women of reproductive age (12-45 years old) and is thought to be one of the leading causes of the female subfertility

* The aim of this work is to study the effect of metformin use for reducing early pregnancy loss in pregnant patients with PCOS
* Research question:

In pregnant women with PCOS, does metformin use decreases the rate of early pregnancy loss?

-Research hypothesis: In Pregnant women with PCOS, metformin may reduce the rate of early pregnancy loss.

ELIGIBILITY:
Inclusion Criteria:

* Age : 25 - 35.
* Pregnant patients in their 1st trimester with history of infertility due to PCOS confirmed by at least 2 of the following criteria ( Rotterdam Criteria )

  * At least twelve small follicles 2-9 mm in at least one ovary; diagnosed by ultra sound examination.
  * Symptoms or biochemical evidence of hyperandrogenism; diagnosed by examination and laboratory investigations.
  * Anovulation or oligo-ovulation with fewer than nine menstrual periods every 12 months : diagnosed by thorough history taking.
* Non diabetic patients who received metformin along with other ovulation-inducing drugs prior to pregnancy.

Exclusion Criteria:

* patients with other causes of infertility other than PCOS
* contraindications to metformin : liver impairment , renal failure.
* Patients with PCOS who didn't receive Metformin with drugs of induction of ovulation before pregnancy.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M kotb, MD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin Arm | Control Arm
Started | 85 | 85
Completed | 83 | 83
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin Arm | Control Arm | Total
Number analyzed (Participants) | 83 | 83 | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 83 | 83 | 166
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (1.6) | 30.1 (1.9) | 30.1 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 83 | 166
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 83 | 83 | 166

OUTCOME MEASURES:

1. Primary Outcome: Miscarriage Rate
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Metformin Arm | Control Arm
Number analyzed (Participants) | 83 | 83
participants | 9 [4.1 to 17.5] | 35 [31.6 to 52.8]

ADVERSE EVENTS:
Arm/Group | Metformin Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/83
Other Adverse Events (participants affected / at risk) | 16/83 | 6/83
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin Arm (N=83) | Control Arm (N=83)
vomiting (Gastrointestinal disorders) | 16 (16) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less